CLINICAL TRIAL: NCT00557128
Title: A Randomized, Open-label, Single-dose, 3-period Crossover Study to Assess the Effect of Food on the Pharmacokinetics of the Final Fixed Dose Combination Formulation of COREG CR and Lisinopril in the Fed and Fasted State.
Brief Title: Study to Examine the Effect of Food on the Pharmacokinetics of the Fixed Dose Combination of COREG CR and Lisinopril.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CFD108410
Record Dates: First submitted 2007-10-24; First posted 2007-11-12 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension
Keywords: COREG CR,; lisinopril,; hypertension,; dose proportionality,; fixed dose combination (FDC)
MeSH Terms: conditions — Hypertension | interventions — Carvedilol; Lisinopril

INTERVENTIONS:
Drug: COREG CR and lisinopril (FDC)

SUMMARY:
This is a randomized, open-label, single-dose, period-balanced, three-period crossover study conducted in healthy subjects designed to evaluate whether the absorption of the FDC formulation is affected by the ingestion of a high fat meal or is altered when taken in a fasted state.

ELIGIBILITY:
Inclusion criteria:

* Healthy volunteer Adult males and females of non-child bearing potential who are between 18 to 55 years of age, inclusively
* Body weight > 60 kg (132 lbs) and body mass index (BMI) between 19 and 33

Exclusion criteria:

* Any clinically relevant abnormality identified on the screening history, physical or laboratory examination, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study.
* Subjects who metabolize carvedilol poorly based on CYP2D6 genotyping as determined at screening.
* Treatment with any prescription or non-prescription drugs (including vitamins, herbal and dietary supplements, as well as grapefruit-containing products) within 7 days or 5 half-lives (whichever is longer) prior to first dose of study medication and until the end of the study. Treatment with any CYP2D6 inhibitors such as but not limited to quinidine, fluoxetine, paroxetine, duloxetine, and terbinofine at least 14 days or 5 half-lives (whichever is longer) prior to Day 1 of Session 1 and until the end of the study.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding Day 1 of Session 1
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Positive urine drug screen (UDS) including alcohol at screening. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Urine Na/creatinine ratio < 0.08 meq/mg.
* Positive for Hepatitis B surface antigen, or HIV.
* Women of child-bearing potential.
* NOTE: Pre-menopausal females with a documented tubal ligation or hysterectomy are eligible. Postmenopausal females are eligible, defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Resting heart rate of ≤ 50 beats per minute (bpm) at screening.
* Any of the following abnormalities on 12-lead ECG during screening:

  * conduction abnormalities denoted by any of the following:
  * PR interval < 120 msec or > 200 msec
  * non-specific IVCD (intra-ventricular conduction delay) with QRS duration ≥ 110 msec and where the morphology does NOT meet criteria for left (LBBB) or right bundle branch block (RBBB)
  * incomplete RBBB as defined by QRS duration ≥100 msec but < 120 msec with RBBB pattern
  * Complete RBBB or LBBB
  * evidence of second- or third- degree AV block
  * pathological Q-waves (Q-wave wider than 0.04 sec or depth greater than 0.4-0.5 mV)
  * evidence of ventricular pre-excitation
  * evidence of left axis deviation (left axis deviation is -30 to -90 degrees) but not normal leftward axis, ST-T wave abnormalities, left bundle branch block and/or right bundle branch block
  * QTcB interval > 450 msec
* Documented history of low blood pressure (average SBP ≤ 110 mm Hg and/or DBP ≤ 50 mm Hg) or blood pressure below these values at time of screening.
* Orthostatic hypotension diagnosed at screening (orthostatic hypotension will be defined as a reduction in systolic blood pressure of 20 mmHg or more and/or a reduction in diastolic blood pressure of 10 mmHg or more for standing vs. supine measurements.
* Donation of blood in excess of 500 mL within a 56-day period including the estimated 442 mL of blood to be drawn during this study.
* History of asthma, COPD and/or hypersensitivity to β-adrenergic blocking agents.
* History of sensitivity to heparin, heparin-induced thrombocytopenia, or sensitivity to any of the study medications or components thereof.
* History of anaphylaxis or anaphalactoid reactions or severe allergic responses to drugs.
* History of angioedema.
* History of sensitivity to carvedilol, lisinopril, alpha-blockers, beta-blockers or ACE inhibitors.
* Unwillingness or inability to follow the procedures outlined in the protocol or inability to provide written informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The effect of food on PK after high fat and standard meal Blood sampling over a 72 hour period post dose in all dosing sessions | 72 hour period post dose in all dosing sessions

SECONDARY OUTCOMES:
Food effect on PK over 72 hours after meals compared to fasting, safety and tolerability assessed by spontaneous Adverse Event reporting, nurse/physician observations, vital sign assessment, ECGs, and clinical labs over 3 session crossover | 72 hours after meals
Other pertinent pharmacokinetic parameters of carvedilol and lisinopril, as data permit, such as Tmax and t1/2 of carvedilol and Tmax and t1/2 of lisinopril

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States